CLINICAL TRIAL: NCT06960824
Title: Real-word Study of the de NOVO Use of Once-daily Extended-release tacrolimuS (LCPT) in Kidney Transplantation Using an ARTificial Intelligence Prognostic System: a Multicenter Prospective Ob-servational Study
Brief Title: Real-word Study of the de NOVO Extended-release tacrolimuS in Kidney Transplantation Using an ARTificial Intelligence
Acronym: NOVOSTART
Status: Not yet recruiting | Type: Observational
Sponsor: Chiesi SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025-A00256-43
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Chronic Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort of patients treated: Cohort of patients treated with Life-Cycle Pharma Tacrolimus-based immunosuppression: Our single-arm study addresses the primary objective.
  Interventions: Drug: Life-Cycle Pharma Tacrolimus; Procedure: Kidney transplantation
- Reference cohort for transplants: Cohorts Transplant reference: two control groups (Tacrolimus twice daily (IR-Tac) and Tacrolimus once daily (ER-Tac)) to determine the main secondary objective.
  Interventions: Procedure: Kidney transplantation

INTERVENTIONS:
Drug: Life-Cycle Pharma Tacrolimus — Patients receiving LCPT Envarsus® [Life-Cycle Pharma Tacrolimus] within 24 hours of kidney transplantation in a once-daily formulation at the discretion of the investiga-tor and in compliance with the summary of product characteristics (SmPC).
  Groups: Cohort of patients treated
Procedure: Kidney transplantation — Kidney transplant patients using the iBox prognostic system (risk prediction system for kidney transplants)

SUMMARY:
The purpose of this study is to assess the clinical efficacy of the LCPT En-varsus [Life-Cycle Pharma Tacrolimus] initiated in de novo (Day 0 of transplantation) using the Biopsy Proven Acute Re-jection and iBox (full and abbreviated algo-rithms).

DETAILED DESCRIPTION:
NovoStart is a descriptive study, prospective, multicenter, real-world evidence de-signed to evaluate the clinical efficacy and safety of Once-Daily Extended-Release Tacroli-mus in kidney transplantation using the iBox prognostic system.

The NovoStart study will be conducted at 13 academic hospitals in France performing kidney transplants.

The study population will comprise three cohorts of patients:

* Cohort of patients treated with Life-Cycle Pharma Tacrolimus-based immunosuppression: Our single-arm study addresses the primary objective.
* Cohorts Transplant reference: two control groups (Twice-Daily Tacrolimus and Once-Daily Tac-rolimus) to determine the main secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* Kidney recipients aged 18 years and older.
* Kidney recipients were transplanted from living or deceased donors
* Patients receiving Envarsus® [Life-Cycle Pharma Tacrolimus] within 24 hours of kidney transplantation in a once-daily formulation at the discretion of the investiga-tor and in compliance with the summary of product characteristics.
* Patients are willing to participate in the study and do not oppose the use of their data.
* Patients are either affiliated with or beneficiaries of a social security scheme.

Exclusion Criteria:

* Contraindications to the use of Life-Cycle Pharma Tacrolimus (Envarsus®).
* Pre-transplant desensitization.
* ABO is incompatible with a living donor.
* Combined transplant (e.g. kidney-heart transplant, kidney-liver transplant).
* Previous bariatric (or bypass) surgery.
* Gastrointestinal problems are likely to affect the absorption of the Life-Cycle Pharma Tacrolimus (Envarsus®).
* Diagnosis of Parkinson's disease or any other neurological syndrome causing tremor.
* Patients who are part of another clinical trial or in a period of exclusion from another clinical trial with a molecule under study.
* Pregnant women or breastfeeding.
* Patients under legal protection (guardianship, curatorship) or deprived of their liberty through judicial or administrative decisions.
* Patients under State Medical Assistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Cohort of patients treated with LCPT-based immunosuppression : we will recruit all kidney recipients aged 18 years and older, regardless of gender, who have received Life-Cycle Pharma Tacrolimus (Envarsus®) once daily within 24 hours of transplantation, as judged by the investigator, and who meet the eligibility criteria.
  2. Reference transplant cohort : The reference transplant cohort is composed of kidney transplant patients from four French centres (Necker, Saint-Louis, Foch and Toulouse hospitals), comprising 4,000 consecutive patients transplanted between 2005 and 2014.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Biopsy Proven Acute Rejection | 12 months
  The primary endpoint is the incidence of Biopsy Proven Acute Rejection between the Life-Cycle Pharma Tacrolimus cohort and the control groups of the transplant reference cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GATAULT, MD, Principal Investigator — CHRU TOURS
Locations (1):
- Chru Tours, Tours, France